CLINICAL TRIAL: NCT01973517
Title: 7T MRI Ferumoxytol-Enhanced Characterization of Multiple Sclerosis and Demyelinating Diseases
Brief Title: High-Field MRI Iron-Based Contrast-Enhanced Characterization of Multiple Sclerosis and Demyelinating Diseases
Status: Withdrawn | Type: Observational
Why Stopped: Logistical factors affecting recruitment
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Zeineh, Protocol Director, Stanford University
Other Study IDs: 27423-001
Record Dates: First submitted 2013-10-16; First posted 2013-10-31 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; MRI; USPIO; Ferumoxytol; Feraheme
MeSH Terms: conditions — Multiple Sclerosis | interventions — Ferrosoferric Oxide; Gadolinium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relapsing Remitting MS: Patients with relapsing remitting multiple sclerosis will be imaged under high-field (7T) MRI prior to and following administration of gadolinium-based contrast (0.1 mmol/kg IV). Afterwards, they will be administered Feraheme 5mg/kg IV via slow push, and they will return 24 hours or later after pharmaceutical administration for post-Feraheme MR imaging.
  Interventions: Drug: Feraheme; Drug: Gadolinium-based contrast

INTERVENTIONS:
Drug: Feraheme — Patients with relapsing remitting multiple sclerosis will be administered Feraheme 5mg/kg IV via slow push once and imaged under high-field MRI at least 24 hours following administration, to allow for adequate clearance of intravascular pharmaceutical.
  Other Names: Ferumoxytol
Drug: Gadolinium-based contrast — Patients with relapsing remitting multiple sclerosis will be administered gadolinium-based contrast at a dose of 0.1 mmol/kg IV once and imaged under high-field MRI immediately following administration.
  Other Names: Gadolinium

SUMMARY:
Feraheme (ferumoxytol) is FDA-approved for iron supplementation and is composed of iron oxide nanoparticles classified among the ultra-small superparamagnetic iron oxides (USPIO). In this project we hypothesize that Feraheme could become a sensitive and specific marker of active inflammation in multiple sclerosis. We will explore this hypothesis taking advantage of ultra high field strength (7T) MRI to further increase the effectiveness of the contrast agent Feraheme at revealing inflammatory activity.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a neurological disorder that affects young adults world-wide. Feraheme (ferumoxytol) is FDA-approved for iron supplementation and is composed of iron oxide nanoparticles classified among the ultra-small superparamagnetic iron oxides (USPIO). After IV injection, the particles are taken up by the monocyte-macrophage system and can also be used to track macrophage infiltration by magnetic resonance imaging (MRI) after systemic injection owing to the strong image contrast of the iron-loaded macrophages. Approximately 24 hours after their IV injection, free particles are cleared from the circulation and MR signal alterations are thought to arise from the capture of particles by circulating phagocytic cells that are attracted to inflammatory lesions.

In this project we hypothesize that Feraheme could become a sensitive and specific marker of active inflammation in multiple sclerosis. We will explore this hypothesis by taking advantage of ultra high field strength (7T) MRI to further increase the effectiveness of the contrast agent Feraheme at revealing inflammatory activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are at least 18 years old and meet the revised diagnostic criteria for multiple sclerosis, relapsing remitting type.
* Patients will be included based on MR evidence of disease activity after Gadolinium (enhanced lesion) on a previous screening MR in the previous 3 weeks days before Feraheme administration.

Exclusion Criteria:

* Children (age < 18)
* Those who lack decision-making capability
* Contraindication to MRI such as pacemaker, other MR-incompatible metal implants or claustrophobia
* Known allergy to dextran or drugs containing iron salts or any previous history of severe allergic reactions
* Evidence of iron overload such as hemochromatosis or other hematologic disorders that imply iron level superior to the normal level.
* Pregnancy or breast feeding.
* History of renal disease or estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) <40ml/min/1.73m?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be composed of patients with the diagnosis of relapsing remitting multiple sclerosis (MS) who are followed at the Stanford Neurosciences Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number and location of enhancing brain lesions seen on 7 tesla MRI following Feraheme administration. | Baseline
  Magnetic resonance images of the brains of subjects will be evaluated independently by two expert readers blinded to the demographic and clinical data. The location and number of multiple sclerosis lesions that enhance following Feraheme administration will be recorded. These lesions will be compared with non-enhancing lesions and lesions that enhance with gadolinium-based contrast.

SECONDARY OUTCOMES:
Number and location of enhancing brain lesions seen on 7 tesla MRI following gadolinium-based contrast administration. | Baseline
  Magnetic resonance images of the brains of subjects will be evaluated independently by two expert readers blinded to the demographic and clinical data. The location and number of multiple sclerosis lesions that enhance following gadolinium-based contrast administration will be recorded. These lesions will be compared with non-enhancing lesions and lesions that enhance with Ferahame.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zeineh, MD, PhD, Study Director — Stanford University; Brian Rutt, PhD, Study Director — Stanford University
Locations (2):
- United States (2):
  - Richard M. Lucas Center for Imaging (of Stanford University), Stanford, California
  - Stanford Hospitals and Clinics, Stanford, California

REFERENCES:
- [Background] Dousset V, Brochet B, Deloire MS, Lagoarde L, Barroso B, Caille JM, Petry KG. MR imaging of relapsing multiple sclerosis patients using ultra-small-particle iron oxide and compared with gadolinium. AJNR Am J Neuroradiol. 2006 May;27(5):1000-5. PMID 16687532
- [Background] Vellinga MM, Oude Engberink RD, Seewann A, Pouwels PJ, Wattjes MP, van der Pol SM, Pering C, Polman CH, de Vries HE, Geurts JJ, Barkhof F. Pluriformity of inflammation in multiple sclerosis shown by ultra-small iron oxide particle enhancement. Brain. 2008 Mar;131(Pt 3):800-7. doi: 10.1093/brain/awn009. Epub 2008 Feb 1. PMID 18245785
- [Background] Tourdias T, Roggerone S, Filippi M, Kanagaki M, Rovaris M, Miller DH, Petry KG, Brochet B, Pruvo JP, Radue EW, Dousset V. Assessment of disease activity in multiple sclerosis phenotypes with combined gadolinium- and superparamagnetic iron oxide-enhanced MR imaging. Radiology. 2012 Jul;264(1):225-33. doi: 10.1148/radiol.12111416. PMID 22723563
- [Background] Daldrup-Link HE, Rydland J, Helbich TH, Bjornerud A, Turetschek K, Kvistad KA, Kaindl E, Link TM, Staudacher K, Shames D, Brasch RC, Haraldseth O, Rummeny EJ. Quantification of breast tumor microvascular permeability with feruglose-enhanced MR imaging: initial phase II multicenter trial. Radiology. 2003 Dec;229(3):885-92. doi: 10.1148/radiol.2293021045. Epub 2003 Oct 23. PMID 14576446
- [Background] Metz S, Lohr S, Settles M, Beer A, Woertler K, Rummeny EJ, Daldrup-Link HE. Ferumoxtran-10-enhanced MR imaging of the bone marrow before and after conditioning therapy in patients with non-Hodgkin lymphomas. Eur Radiol. 2006 Mar;16(3):598-607. doi: 10.1007/s00330-005-0045-9. Epub 2005 Nov 12. PMID 16284770
- [Background] Pai AB, Nielsen JC, Kausz A, Miller P, Owen JS. Plasma pharmacokinetics of two consecutive doses of ferumoxytol in healthy subjects. Clin Pharmacol Ther. 2010 Aug;88(2):237-42. doi: 10.1038/clpt.2010.80. Epub 2010 Jun 30. PMID 20592725
- [Background] Provenzano R, Schiller B, Rao M, Coyne D, Brenner L, Pereira BJ. Ferumoxytol as an intravenous iron replacement therapy in hemodialysis patients. Clin J Am Soc Nephrol. 2009 Feb;4(2):386-93. doi: 10.2215/CJN.02840608. Epub 2009 Jan 28. PMID 19176796
- [Background] Schwenk MH. Ferumoxytol: a new intravenous iron preparation for the treatment of iron deficiency anemia in patients with chronic kidney disease. Pharmacotherapy. 2010 Jan;30(1):70-9. doi: 10.1592/phco.30.1.70. PMID 20030475
- [Background] Lu M, Cohen MH, Rieves D, Pazdur R. FDA report: Ferumoxytol for intravenous iron therapy in adult patients with chronic kidney disease. Am J Hematol. 2010 May;85(5):315-9. doi: 10.1002/ajh.21656. PMID 20201089
- [Background] Dousset V, Delalande C, Ballarino L, Quesson B, Seilhan D, Coussemacq M, Thiaudiere E, Brochet B, Canioni P, Caille JM. In vivo macrophage activity imaging in the central nervous system detected by magnetic resonance. Magn Reson Med. 1999 Feb;41(2):329-33. doi: 10.1002/(sici)1522-2594(199902)41:23.0.co;2-z. PMID 10080281
- [Background] Dousset V, Ballarino L, Delalande C, Coussemacq M, Canioni P, Petry KG, Caille JM. Comparison of ultrasmall particles of iron oxide (USPIO)-enhanced T2-weighted, conventional T2-weighted, and gadolinium-enhanced T1-weighted MR images in rats with experimental autoimmune encephalomyelitis. AJNR Am J Neuroradiol. 1999 Feb;20(2):223-7. PMID 10094342
- [Background] Floris S, Blezer EL, Schreibelt G, Dopp E, van der Pol SM, Schadee-Eestermans IL, Nicolay K, Dijkstra CD, de Vries HE. Blood-brain barrier permeability and monocyte infiltration in experimental allergic encephalomyelitis: a quantitative MRI study. Brain. 2004 Mar;127(Pt 3):616-27. doi: 10.1093/brain/awh068. Epub 2003 Dec 22. PMID 14691063
- [Background] Ladewig G, Jestaedt L, Misselwitz B, Solymosi L, Toyka K, Bendszus M, Stoll G. Spatial diversity of blood-brain barrier alteration and macrophage invasion in experimental autoimmune encephalomyelitis: a comparative MRI study. Exp Neurol. 2009 Nov;220(1):207-11. doi: 10.1016/j.expneurol.2009.08.027. Epub 2009 Sep 4. PMID 19733560
- [Background] Chin CL, Pai M, Bousquet PF, Schwartz AJ, O'Connor EM, Nelson CM, Hradil VP, Cox BF, McRae BL, Fox GB. Distinct spatiotemporal pattern of CNS lesions revealed by USPIO-enhanced MRI in MOG-induced EAE rats implicates the involvement of spino-olivocerebellar pathways. J Neuroimmunol. 2009 Jun 25;211(1-2):49-55. doi: 10.1016/j.jneuroim.2009.03.012. Epub 2009 Apr 5. PMID 19346009
- [Background] Petry KG, Boiziau C, Dousset V, Brochet B. Magnetic resonance imaging of human brain macrophage infiltration. Neurotherapeutics. 2007 Jul;4(3):434-42. doi: 10.1016/j.nurt.2007.05.005. PMID 17599709